CLINICAL TRIAL: NCT04682171
Title: Effects of Low Level Laser Therapy on Knee Pain and Function in Patients With Knee Osteoarthritis
Brief Title: Low Level Laser Therapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1040 Abeel Ashraf
Record Dates: First submitted 2020-12-21; First posted 2020-12-23 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee pain; Knee function; Degenerative knee disease
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level Laser Therapy (Experimental): Low Level Laser Therapy and Conventional Exercise therapy
  Interventions: Other: Low level laser therapy; Other: Conventional Exercise Therapy
- Conventional ExerciseTherapy (Active Comparator): Conventional ExerciseTherapy
  Interventions: Other: Conventional Exercise Therapy

INTERVENTIONS:
Other: Low level laser therapy — * Gallium aluminium arsenide laser device will be used with wavelength of 850nm, power 100 mW, spot size of 1.0 mm and energy of 6J/point for 60seconds. Total 8 points will be irradiated. It will take 20 minutes.
  * Patient will receive treatment in supine position with the affected knee(s) slightly flexed supported by the pillow or rolled towel.
  * On the affected knee the laser probe will placed with full contact with skin at 8 points. Three points at medial side of the knee, three points at lateral side and two points at the medial edge of the bicep femoris muscle tendon and semitendinosus muscle tendon in the popliteal fossa
  Arms: Low level Laser Therapy
Other: Conventional Exercise Therapy — 1. Quadriceps isometric strengthening exercises.
  2. Range of motion and active stretching exercises applied to hamstring and quadriceps muscle.
  3. Hamstring muscle isometric exercises
  4. Active ankle pump.
  5. Short arc terminal extension exercises for the knee joint.
  6. Static and dynamic strengthening exercises for the hip abductors, adductors and extensor group of muscles.
  7. Non-weight bearing progressive resistance exercises with weighted cuffs, with progression to closed chain exercises as patient's pain allows.
  8. Isometric exercises were applied with 6 second contractions and rest period of 2 seconds. Isotonic exercises were started as 10 repetitions with half of weight of 10 RM, 10 repetitions with three fourth of this weight and 10 repetitions with whole 10 RM

SUMMARY:
The study will be Randomized Controlled Trial. It will be conducted in Allied Hospital Faisalabad. The study will be completed in four months duration. Consecutive sampling technique will be used for data collection. A sample size of 40 patients will be taken in this study. Participants will be divided into two groups. Group A will be treated by LLLT and conventional exercises. Group B will perform conventional exercises only. Numeric Pain Rating Scale will be used to measure pain. Western Ontario McMaster Universities Osteoarthritis Index Score (WOMAC) and Sit to stand test will be used to measure knee function. Goniometry will be used to measure ROM of knee. The participants will fill numeric pain rating scale and WOMAC as subjective measurements. Knee flexion ROM will be measured with universal Goniometer. Total 12 sessions will be given with three sessions per week. Post treatment readings will be taken at the end of 4th week. Data will be analyzed on SPSS 25.

DETAILED DESCRIPTION:
One of the most common forms of arthritis is Osteoarthritis. Approximately 15% of the population is affected by the disease. The prevalence of the disease increases with the age, with the peak incidence at fourth decade of life. Study shows that in Southern Pakistan mean age of the patients suffering from Osteoarthritis was 58 years. The disease was more dominant in women with the 3:8 male to female ratio. Study shows that 13.9% of adults aged 25 years and above and 33.6% of older adults aged over 65 years are suffering from osteoarthritis.

According to Johnston County Osteoarthritis Project prevalence of symptomatic knee OA was recorded to be 16% and 28% for radiographic knee OA. Kellgren-Lawrence classified knee osteoarthritis based on the appearance of osteophytes in knee AP radiographs. Grades 0-4 were assigned with >2 indicating radiographic OA. Pain and stiffness are significant clinical features of OA which leads to reduced physical function while articular cartilage degeneration is considered to be important pathological feature of OA. Genetic factors, age-related physiological changes and biomechanical factors are considered risk factors of osteoarthritis. Several studies shows that increased age and BMI increases the risk of knee osteoarthritis. One of the important factors in knee osteoarthritis is being overweight.Physical inactivity is also associated with osteoarthritis. Most notable symptom of osteoarthritis is pain which is also determining factor of disability in patients with osteoarthritis. Pain increases physical inactivity which leads to increased body weight and eventually predispose the person to osteoarthritis.Quadriceps weakness may contribute to prompt clinical finding of knee osteoarthritis. Pain of osteoarthritis may causes reduced quadriceps strength. However some studies reveal that quadriceps weakness plays as a risk factor for knee osteoarthritis especially in females. Reduced muscle strength was reported in 24% of patients with Kellgren-Lawrence grade II knee OA. It is widely accepted that among the patients with knee osteoarthritis quadriceps weakness is caused by muscle atrophy which reduces muscle strength. It is reported that age-related quadriceps weakness is linked with functional limitations and increased rate of falling among elders.

Treatment options for osteoarthritis include pharmacological and non-pharmacological methods. The primary goal of these treatments is to relieve joint pain and improve functional quality of life. Non-steroidal anti inflammatory (NSAIDS) are used widely but their use is now limited due

to high frequency of side effects specially side effects of gastrointestinal tracts.Therefore non-pharmacological treatment is preferred for elderly patients. Non-pharmacological treatment includes weight reduction, manual therapy, strengthening exercises, electrical stimulation, ultrasound, interferential current and laser therapy.

Low level laser therapy (LLLT) is non-invasive and painless modality used for the treatment of knee osteoarthritis. Studies show that it markedly alleviates both acute and chronic conditions such as carpal tunnel syndrome, knee injuries, low back pain, chronic arthritis and rheumatoid arthritis. Due to its stimulatory effect on tissue metabolism and ability to regulate the inflammatory effect after knee injuries, LLLT is considered as a favorable therapeutic modality for OA. It is reported that LLLT was effective for fibroblast and osteoblast proliferation, bone regeneration, collagen synthesis, cellular oxygenation and release of neurotransmitters linked with pain modulation.

Evidence shows that regular physical activity reduces pain and improves physical function among the patients with knee OA. However being inactive and disuse of affected limb may disturbs joint mechanics leading to softening of articular cartilage which leads to rapid degeneration of cartilage. This study will focus on additive effects of LLL therapy on knee OA patients for improving pain and function. This study will provide an insight in traditional methods that are used in OA patients.

3. LITERATURE REVIEW: Osteoarthritis is the most common form arthritis which is overall ranked among 50 common sequelae of injuries and diseases. Almost 250 million people or 4% of the world's population is affected by osteoarthritis. It is generally divided into primary OA and secondary OA. Etiology of primary OA is not clear but some factors such as genetic factor, ethnicity, age related changes and biomechanical factors play an important role. Post traumatic, dysplastic, infectious, inflammatory or biomechanical etiologies are common cause of secondary OA.

Females are more affected with hand, feet and knee OA. Women are more subjected to severe knee OA than men especially after menopause due to the role of estrogen. Oestrogen unmasks the symptoms of OA by increasing pain sensitivity(1). According to a study male to female ratio affected by OA in Pakistan is 3:8.

Most significant symptom of knee OA is pain leading to increased physical inactivity which increases body weight and predispose the person to OA. Obesity is also a risk factor for developing knee OA.

Pain in knee OA also reduces strength in quadriceps muscle. Quadriceps weakness in OA may be associated with the action of quadriceps during gait. Shock absorption at the knee is provided by eccentric contraction of quadriceps. The spontaneous loading at the knee resulting from inability to compensate the large compressive forces leads to quadriceps weakness and osteoarthritic changes.

A number of evidence shows that exercise reduces the symptoms of OA and improves the knee joint function. However the most advantageous type or combination of exercises is uncertain. Physical inactivity and disuse of the affected limb result in loss of flexibility around knee joint leading to impaired joint mechanics and increased clinical findings of pain. Participation in physical activity and exercise has been recorded to improve joint function and beneficial for the treatment of knee OA.

Physical therapy interventions for knee OA include electrical stimulation, manual therapy, strengthening exercises, ultrasound, interferential current therapy, laser therapy and orthotic devices. Low level laser therapy (LLLT) has been widely used for relieving pain in many

musculoskeletal disorders. It has been considered as non-invasive and safe treatment for knee OA due its stimulatory effect on tissue metabolism and ability to regulate inflammatory process after injury Osteoarthritis is more common in females as compared to males. Pain, joint stiffness and reduced physical activity are prominent symptoms of knee OA. Genetic factors, reduced BMI, overweight, age related physical changes and quadriceps weakness are considered risk factors for knee OA. Physical inactivity disturbs the knee biomechanics and increases the symptoms of knee OA. Studies show that exercise helps to improve the symptoms of knee OA and enhance physical function. Low level laser therapy is non-invasive and painless therapeutic modality used for treating knee OA. Evidence proves that LLLT helps in relieving pain of OA and improving microcirculation due to its stimulatory effect on tissue metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* Patients with age 45-65 years
* Patients with knee OA of grade II or III according to Kellgren-Lawrence grade.
* Pain intensity ranging between> 5 measured by Numeric Pain Rating Scale.
* Patients who had minimum score of 25 on the Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) total score.
* Patients having knee pain for at least 3 months.

Exclusion Criteria:

* Patients with pain in other lower limb joints.
* Patients with symptomatic hip osteoarthritis.
* Patients with knee surgery in last 6 months.
* Patients with complaint of cancer, diabetes, neurological deficit or uncontrolled hypertension

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  NPRS is a segmented version of Visual Analogue Scale (VAS). It consists of number from 0 to 10. Patient selects a number that best reflects his/her pain intensity where 0 is no pain and 10 is maximum pain. For construct validity, NPRS was highly correlated to Visual Analogue Scale (VAS) (0.86-0.95).The test-retest reliability of this scale is recorded to be 0.96
Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | 4th week
  WOMAC is a valid and reliable outcome measuring tool for evaluating patients with hip and knee osteoarthritis. It measures degree of pain (5 questions), severity of joint stiffness (2 questions) and physical functions (17 questions). WOMAC score was recorded on five points Likert Scale ranging from 0-4 where 0 shows no pain/limitation and 4 shows extreme pain/limitation. Maximum score for pain, joint stiffness and physical function are 28, 8 and 68 respectively with total of 96 scores indicating severe disease.

SECONDARY OUTCOMES:
Knee Rang of Motion (Flexion and Extension) | 4th Week
  Universal goniometer is a valid and reliable tool for measuring knee range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Allied Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson VL, Hunter DJ. The epidemiology of osteoarthritis. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):5-15. doi: 10.1016/j.berh.2014.01.004. PMID 24792942
- [Background] Alghadir A, Omar MT, Al-Askar AB, Al-Muteri NK. Effect of low-level laser therapy in patients with chronic knee osteoarthritis: a single-blinded randomized clinical study. Lasers Med Sci. 2014 Mar;29(2):749-55. doi: 10.1007/s10103-013-1393-3. Epub 2013 Aug 3. PMID 23912778
- [Background] Akhter E, Bilal S, Kiani A, Haque U. Prevalence of arthritis in India and Pakistan: a review. Rheumatol Int. 2011 Jul;31(7):849-55. doi: 10.1007/s00296-011-1820-3. Epub 2011 Feb 18. PMID 21331574
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Jackson BD, Wluka AE, Teichtahl AJ, Morris ME, Cicuttini FM. Reviewing knee osteoarthritis--a biomechanical perspective. J Sci Med Sport. 2004 Sep;7(3):347-57. doi: 10.1016/s1440-2440(04)80030-6. PMID 15518300
- [Background] Jarvholm B, Lewold S, Malchau H, Vingard E. Age, bodyweight, smoking habits and the risk of severe osteoarthritis in the hip and knee in men. Eur J Epidemiol. 2005;20(6):537-42. doi: 10.1007/s10654-005-4263-x. PMID 16121763
- [Background] Christensen R, Bartels EM, Astrup A, Bliddal H. Effect of weight reduction in obese patients diagnosed with knee osteoarthritis: a systematic review and meta-analysis. Ann Rheum Dis. 2007 Apr;66(4):433-9. doi: 10.1136/ard.2006.065904. Epub 2007 Jan 4. PMID 17204567
- [Background] Rosemann T, Kuehlein T, Laux G, Szecsenyi J. Osteoarthritis of the knee and hip: a comparison of factors associated with physical activity. Clin Rheumatol. 2007 Nov;26(11):1811-7. doi: 10.1007/s10067-007-0579-0. Epub 2007 Mar 2. PMID 17332977
- [Background] Huang Z, Chen J, Ma J, Shen B, Pei F, Kraus VB. Effectiveness of low-level laser therapy in patients with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Sep;23(9):1437-1444. doi: 10.1016/j.joca.2015.04.005. Epub 2015 Apr 23. PMID 25914044
- [Background] Alqualo-Costa R, Thome GR, Perracini MR, Liebano RE. Low-level laser therapy and interferential current in patients with knee osteoarthritis: a randomized controlled trial protocol. Pain Manag. 2018 May;8(3):157-166. doi: 10.2217/pmt-2017-0057. Epub 2018 May 3. PMID 29722602
- [Background] Alfredo PP, Bjordal JM, Dreyer SH, Meneses SR, Zaguetti G, Ovanessian V, Fukuda TY, Junior WS, Lopes Martins RA, Casarotto RA, Marques AP. Efficacy of low level laser therapy associated with exercises in knee osteoarthritis: a randomized double-blind study. Clin Rehabil. 2012 Jun;26(6):523-33. doi: 10.1177/0269215511425962. Epub 2011 Dec 14. PMID 22169831
- [Background] Esser S, Bailey A. Effects of exercise and physical activity on knee osteoarthritis. Curr Pain Headache Rep. 2011 Dec;15(6):423-30. doi: 10.1007/s11916-011-0225-z. PMID 21956792